CLINICAL TRIAL: NCT05498415
Title: Sleep Move Stand Study
Brief Title: Feasibility, Acceptability, and Efficacy of the Sleep Move Stand Study
Acronym: SMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Lucas Carr, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201812789
Record Dates: First submitted 2022-07-28; First posted 2022-08-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Physical Inactivity; Sedentary Behavior; Sleep; Cognitive Function
MeSH Terms: conditions — Sedentary Behavior | interventions — Educational Status; Fitness Trackers

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be randomly assigned to group A (control) or group B (treatment) but will not be told which group they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Active Comparator): Participants will receive basic education information on physical activity, sedentary behavior, and sleep for 8 weeks.
  Interventions: Behavioral: Education
- Education + Health Coaching + Activity Monitor (Experimental): Participants will receive education information on physical activity, sedentary behavior and sleep plus health coaching plus a Fitbit activity monitor for 8 weeks.
  Interventions: Behavioral: Education; Behavioral: Health coaching; Behavioral: Activity Monitor

INTERVENTIONS:
Behavioral: Education — Participants will receive standard of care education information on physical activity, sedentary behavior, and sleep via a mobile app for 8 weeks.
Behavioral: Health coaching — Participants will meet with a health coach weekly for 8 weeks
  Arms: Education + Health Coaching + Activity Monitor
Behavioral: Activity Monitor — Participants will receive a Fitbit activity monitor to support goal setting and self monitoring of behaviors.
  Arms: Education + Health Coaching + Activity Monitor

SUMMARY:
The overarching goal for this project is to develop a service-learning program that provides students excellent hands on training and patients with an excellent service that advances their health and well-being. The aim of this study is to test the feasibility, acceptability and efficacy of an 8 week intervention on physical behaviors, cognitive function, and health outcomes compared to a control condition among sedentary, overweight and obese adults.

DETAILED DESCRIPTION:
The overarching goal for this project is to develop and test a service-learning health promotion intervention that provides students hands on training and patients with a service that advances their health and well-being. Inactive but healthy community members and patients being treated at our local hospital will be recruited to participate. Interested volunteers will be randomized into one of two 8 week interventions. The control group will receive basic education information on physical activity, sedentary behavior, and sleep that is consistent with standard of care. These materials will be accessed via a health coaching software program called Healthie. The treatment group will receive the same education information plus health coaching and a Fitbit activity monitor to further support behavior change. Participants will be blinded to their group assignment. Major outcomes include physical activity, sedentary behavior, sleep, cognitive function, and several health outcomes. Success on whether or not the program is found to be feasible, acceptable, and effective.

ELIGIBILITY:
Inclusion Criteria:

* Physically inactive
* Overweight or obese
* Healthy enough to safely engage in regular physical activity

Exclusion Criteria:

* <18 years or >80 years
* Report achieving more than 75 minutes/week of moderate to vigorous intensity physical activity
* Underweight or normal weight (BMI <25.0 mg/kg2)
* Do not intend on becoming more active in the next 3 months
* Not able to commit to a 8 week physical activity program
* No access to smartphone capable of sending and receiving text messages
* Self report mobility issues or diagnosed diseases that prevent safely engaging in regular physical activity
* Planned surgery in the next 12 weeks
* Pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Physical activity | Change from baseline daily steps at 8 weeks
  Daily steps will be measured with an ActivPAL monitor
Sedentary Behavior | Change from baseline daily minutes sedentary at 8 weeks
  Daily minutes spent sedentary will be measured with an ActivPAL monitor
Sleep | Change from baseline daily minutes spent sleeping at 8 weeks
  Daily minutes spent sleeping will be measured with an ActivPAL monitor

SECONDARY OUTCOMES:
Cognitive function | Change from baseline cognitive function at 8 weeks
  Facets of cognitive function will be measured with the NIH Toolbox application

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share IPD with other researchers.